CLINICAL TRIAL: NCT06627907
Title: Hemodynamic Response to the End-expiratory Occlusion Test to Titrate Fluid Challenge in Operating Room.
Acronym: FC_EEOT
Status: Not yet recruiting | Type: Observational
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: FC_EEOT
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Fluid Responsiveness Predictability
Keywords: Fluid challenge; End-expiratory occlusion test; FLuid responsiveness; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Patients receiving a fluid challenge
  Interventions: Other: fluid challenge; Diagnostic Test: end-expiratory occlusion test

INTERVENTIONS:
Other: fluid challenge — The study protocol is started during a period of intraoperative hemodynamic stability, as previously defined (i.e. change in mean arterial pressure of less than 10% during 5 minutes [32, 33]). The study protocol is was the following: 1) a set of measurements was recorded (T0) at a baseline 2) (T1) after one minute the EEOT is then performed by stopping the mechanical ventilation for 30 seconds (T2 - end of the EEOT test); 3) (T3) a FC of overall 6 mL/Kg of crystalloid solution is infused over 10 minutes (T4 end of the FC). The attending anesthetist is allowed to interrupt the protocol at any stage for either hemodynamic instability or any other adverse effects requiring urgent treatment.
  The protocol is entirely intraoperative and data collections ends after FC administration. No follow-up is needed.
  The mentioned timepoints T0 - T1 - T2, corresponding to intrapeortive data recording points are also the endpoints of the study. At each specific timepoint, a marker is added to the M
Diagnostic Test: end-expiratory occlusion test — The study protocol is started during a period of intraoperative hemodynamic stability, as previously defined (i.e. change in mean arterial pressure of less than 10% during 5 minutes [32, 33]). The study protocol is was the following: 1) a set of measurements was recorded (T0) at a baseline 2) (T1) after one minute the EEOT is then performed by stopping the mechanical ventilation for 30 seconds (T2 - end of the EEOT test); 3) (T3) a FC of overall 6 mL/Kg of crystalloid solution is infused over 10 minutes (T4 end of the FC). The attending anesthetist is allowed to interrupt the protocol at any stage for either hemodynamic instability or any other adverse effects requiring urgent treatment.
  The protocol is entirely intraoperative and data collections ends after FC administration. No follow-up is needed.
  The mentioned timepoints T0 - T1 - T2, corresponding to intrapeortive data recording points are also the endpoints of the study. At each specific timepoint, a marker is added to the M

SUMMARY:
Personalzing intraoperative anesthetic fluid management may help in preventing fluid accumulation and related complications.

Fluids are gine as boluses in operating room (the so-called FC). The response to the FC is due to several physiological conditions related to the "preload dependency" (i.e. the intrinsic ability of the heart of increasing the stroke volume - SV - in response to fluid administration).

The minimal volume required to appropriately "challenge" the cardiovascular system is 4 ml/kg of fluid, but higher volumes (up to 6 ml/kg may be needed).

Predicting the response to FC administration may be possible by applying a physiological test (called functional hemodynamic test), such as the end-expiratory occlusion test, consisting in interrupping the mechanical ventilation and hence promoting venous return and consequente SV changes. The percentage of SV increase associated to EEOT may predict fluid responsiveness to the FC (patients responders will increase SV to a bigger extent, as compared to non-responders)

DETAILED DESCRIPTION:
A two-step statistical approach will be used to define the best model to predict the fluid responsiveness.

1. A univariable logistic regression model to test the association of the considered hemodynamic variables provided by the hemodynamic monitoring with the primary outcome (fluid responsiveness at 10th minute). Then a multivariable analysis incorporating the variable in univariable analysis with a p < 0.2, after testing the colinearity and interactions. Significance threshold for multivariable analysis will be set to 0.05
2. A Hosmer and Lemeshow test was calculated to evaluate goodness of fit for the logistic regression model, the Informative criterion metrics, such as Akaike Infromation Criterion, AIC) and the receiver operating characteristic (ROC) curve [standard error, (SE)] analysis evaluated the performance of predictive items for FC response (i.e.Y = dependent variable =SVI increasedby ≥ 10%) 10 minutes (Y10) after FC infusion. The absence of a significant increase in the likelihood value afteromission of each of the remaining variables was checked.

To define the best model to predict the amount of fluid in responder group a machine-learning approach will be considered where Y = dependent variable = total amount of crystalloids to obtained SVI ≥ 10% after FC infusion, X = matrix of parameters. The final model decision will be made among following commonly used regression algorithms: linear reagression, Lasso Regression or Ridge Regression. The model performance assessment will be made using metrics like Mean Squared Error (MSE) or R-squared. K-fold cross-validation technique will be applied to get a more robust estimate of the model's performance.

The hemodynamic values of responders and non-responders at each step of the protocol are analyzed with a one -way analysis of variance for repeated measurements (ANOVA) and Geisser -Greenhouse (G-G) correction as ajustement for lack of sphericity if needed. Post-hoc pairwise multiple comparisons analysis are performed using Tukey's test to control familywise error.

To understand whether hemodynamic changes after EEOT could help in the prediction of minimal dose of FC the study will enroll 2-year evaluable patients, and the final numer will be foreseen in about 300, with aroud 500 fluid challenge.

The sample size will allow us to perform three step:

4. an initial step of 50 patients to understand which variables of hemodynamic changes after EEOT will affect the minimal dose of FC. In this initial part a variable will be considered interesting if the relative p value will be under 0.1 5. A second step including 200 patients' data to create the model, considering also variables interactions 6. A finel step of 50 patients to validate the model

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥ 18 years
2. Scheduled for elective supine abdominal laparotomic or neuro surgery, requiring invasive arterial monitoring and continuous hemodynamic monitoring
3. All the patients must be able to sign an informed consent at the admission

Exclusion Criteria:

1. Any recurrent cardiac arrhythmias
2. Reduced left (ejection fraction <30%) or right (systolic peak velocity of tricuspid annular motion <0.17 m/s) ventricular systolic function
3. Urgent / Emergent surgery
4. Liver surgery
5. Laparoscopic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective abdominal or neuro surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
fluid responsiveness | 10 minutes
  stroke volume index > or equal to 10%